CLINICAL TRIAL: NCT06217770
Title: Retrospective, Non-interventional Study Assessing the Real-Life Use of The Long- Acting Gonadotropin-releasing Hormone Agonist as A Treatment for Locally Advanced or Meta-static Prostate Cancer in Hong Kong.
Brief Title: Retrospective Study to Assess Real-Life Use of The Long Acting GnRH Agonist as Prostate Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Principal Investigator, Chi Fai NG, Professer, Chinese University of Hong Kong
Other Study IDs: CRE-2023.180
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is a retrospective review of the electronic medical record of patients on long-acting triptorelin in Hong Kong.

DETAILED DESCRIPTION:
Prostate cancer is the second most prevalent cancer in men worldwide. Analogues of natural gonadotrophin releasing hormone (GnRH) are currently available in clinical practice to induce castration in subjects with prostate cancer. While 6 month formulation of Triptorelin has been approved since 2018 for controlling tumor growth in subjects with prostate cancer living in Hong Kong, to date, there are no published clinical data regarding the use and efficacy of the 6 month formulation in Chinese subjects with Chinese heritage. To better understand the real-world experience of long-acting GnRH agonist, there is an unmet need for a retrospective, noninterventional review to collect data regarding the use of the long-acting formulation GnRH in clinical practice as a treatment for prostate cancer. The purpose of this study is to collect data on healthcare characteristics and the treatment patterns in the real-world setting, as well as to understand the profile of the subject population using long-acting formulation GnRH agonist.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Chinese heritage
* Prostate cancer patients with the following disease status:

  * High-risk prostate cancer having hormonal therapy as neoadjuvant / adjuvant treatment for prostatectomy or radiotherapy; or
  * Advanced / metastatic prostate cancer treated with long-term hormonal therapy; or
  * After primary therapy (surgery or radiotherapy) with biochemical recurrence; or
  * Castration-resistant prostate cancer status
* Received at least one dose of 6-month Gonadotropin-releasing Hormone Agonist triptorelin formulation
* Having at least 6 months of follow-up after administration of the 3-month to 6-month Gonadotropin-releasing Hormone Agonist triptorelin

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High risk prostate cancer patient of Chinese heritage from Prince of Wales Hospital since 1 Sept 2018.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
The usage pattern of the long-acting Gonadotropin-releasing Hormone Agonist agonist triptorelin in real-life clinical practice | 6 months
  The duration and type of GnRH agonist

SECONDARY OUTCOMES:
The effectiveness of the long-acting Gonadotropin-releasing Hormone Agonist agonist triptorelin in inducing and maintaining castration | 6 months
  It is assessed by the PSA , testosterone level

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rawla P. Epidemiology of Prostate Cancer. World J Oncol. 2019 Apr;10(2):63-89. doi: 10.14740/wjon1191. Epub 2019 Apr 20. PMID 31068988
- [Background] Weckermann D, Harzmann R. Hormone therapy in prostate cancer: LHRH antagonists versus LHRH analogues. Eur Urol. 2004 Sep;46(3):279-83; discussion 283-4. doi: 10.1016/j.eururo.2004.05.006. PMID 15306097